CLINICAL TRIAL: NCT04161521
Title: Conservative Surgical Novel Technique of Placenta Accreta in Menoufia University Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia Obstetrics and Gynecology Group (Other)
Responsible Party: Principal Investigator, Dr Hamed Ellakwa, Professor Hamed Ellakwa, Menoufia Obstetrics and Gynecology Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Menoufia OGG
Record Dates: First submitted 2019-11-05; First posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Placenta Accreta patients (Other): of 60 pregnant female diagnosed as placenta previa accreta recuirted from Obstetrics and Gynecology Department , Menoufia University Hospital.
  Interventions: Procedure: Novel Technique of Placenta Accreta in Menoufia University Hospital

INTERVENTIONS:
Procedure: Novel Technique of Placenta Accreta in Menoufia University Hospital — * Classical CS to decrease haemorrhage from placental bed.
  * Delievery of the fetus.
  * At the delivery 10 UI of oxytocin IV will be injected.
  * The placenta is not attempted to be delievered.
  * Opening of the broad ligament via round ligament division and ligation.
  * Gentle dissection of the urinary bladder from lateral to medial.
  * Bilateral uterine artery clamping at low level below the placental bed .
  * Gentle attempt to deliver The placenta.
  * If the placenta is delievered we will do bilateral uterine artery ligation at multiple levels and multiple square compression sutures(if needed) for proper hemeostasis at the placental bed. Then closure of uterine incision.
  * If the placenta is not delievered we will do segmental ressection of lower uterine segment including the placenta .
  * Intraperitoneal drain insertion.

SUMMARY:
Evaluation of maternal morbidity and mortality of our novel surgical procedure for conservative management of placenta accreta in our tertiary referral institute.

DETAILED DESCRIPTION:
A descripative cohort study which included 60 pregnant women recuirted from Obstetrics and Gynecology Department, Menoufia University Hospital and diagnosed as placenta previa accreta.

• Ethical considerations: Ethics: The study was approved by Ethical Committee of Menoufia Faculty of Medicine.

Consent: after explanation of surgical procedure of the study, an informed written consent was obtained from all cases included in this study.

Sample size: (No= 60) Based on previous studies regarding MAP, The incidence of placenta accreta = 1/2500 , so the calculated sample size for this study was 59 which to be around 60 with confidence level 95% margin of error 5% (Pliskow S et al., 2009).

Inclusion criteria:

1. Age between 20 - 40 years old.
2. Gestational age between 28 - 38 weeks.
3. Any patient diagnosed as placenta previa with ultrasound criteria of accretion.

   * Criteria of accretion by Colour Doppler ultrasound include: (Berkley et al., 2013).

     1. The presence of irregular shaped placental lacunae within the placenta.
     2. Thinning of myometrium overlying the placenta.
     3. Absence of retroplacental 'non-lucent line'.
     4. Protrusion of the placenta into the bladder.
     5. Increased vascularity of the uterine serosa-bladder interface.
     6. Turbulent blood flow through the lacunae on Doppler ultrasonography.
   * All patients were subjected to the following:

I. Detailed history taking:

1. Personal history: name ,age, address, occupation, marietal status, number of children ,age of the youngest child, the gender of the children and special habbits of medical importance like smoking.
2. Past history: past medical history (e.g. diabetes mellitus, hypertension, renal disease, liver disease and any systemic disease like cardiac or pulmonary diseases), past surgical history (any operation done before), blood transfusion, drugs taken and allergy from any drug.
3. Family history: hypertension, diabetes mellitus, consanguinity.
4. Menstrual history: LMP (the first day of last menstrual period), duration, frequency, regularity of period, presence of dysmenorrhea and EDD (the expected date of delivery).
5. Obstetric history : gravidity, parity, number of deliveries, mode of delivery (normal vaginal delivery or cesarean delivery) , place of delivery, the reason for cesarean delivery, any operative complications, number of children and their gender , any neonatal complications, number of abortions, gestational age of them, if abortion followed by surgery like evacuation and curettage.

II. Clinical examination:

1. General examination:

   * General condition.
   * Vital signs including blood pressure, pulse, temperature.
   * Height, weight and body mass index (BMI).
   * Neck : thyroid gland, neck veins and pulsations.
   * Chest : lung, heart, breasts.
   * Upper and lower limbs (edema , varicosities).
2. Abdominal examination :

   1. Inspection :

      Size, shape, pigmentation (linea nigra),stria gravidarum and scars (like cesarean section scars).
   2. Palpation:

      To detect tenderness, rigidity and fundal level.
   3. Auscultation:

      Fetal heart sounds.

      III. Investigations :
      * Preoperative labaratory investigations like complete blood count (CBC), prothrombin time (PT), liver function, kidney function, virology and ECG.
      * Obstetric ultrasound:

      Fetal observation : transabdominal pelvic ultrasound was performed to detect fetal presentation, lie, viability ( by observation of fetal heart movement), gestational age by measuring biparital diameter, femur length and abdominal circumference) and fetal weight.

      Placenta observation : site (anterior or posterior), position in realtion to internal os to determine type of placenta previa and colour Doppler to determine grade of accretion ( accrete, increta, percreta and focal aacretion) and criteria of accretion.

      Surgical Procedure:

      Uterine conservation required multidisciplinary team including the obstetrician, anasethetist and urologist in certain cases.
      1. Preoperative prophylactic antibiotic was given to study cases prior to skin incision tio avoid postoperative endometritis in the form of 2gm ampicillin. (ACOG, 2011)
      2. Preoperative blood cross matching as availability of adequate blood was mandatory.
      3. Operative Steps:

         * Elective CS at 36 weeks to 37 weeks was done.
         * Prior to delivery, two large bore venous lines were placed.
         * General anasethia was recommended.
         * Foley catheter was inserted.
         * Sterilization by povidone- iodine scrub and toweling.
         * Midline incision was done as it made field obvious.
         * Incision of subcutaneous tissue and rectus sheath.
         * Separation of two recti.
         * Classical CS (vertical incision in the upper uterine segment) or high transverse uterine incision was done to decrease haemorrhage through placental bed and to avoid urinary bladder injury as it may be adherent to lower uterine segment in some cases.
         * Delievery of the fetus by gental fundal pressure.
         * At the delivery of the fetus 10 UI of oxytocin IV was injected to help uterus to contract and avoid postpartum atony and to decrease blood loss during delivery.
         * No attempt to the deliver the placenta
         * Exteriorization of uterus including placenta clamped.
         * Two corners of the uterine incision, and the superior and inferior lips, were clamped immediately by four clamps.
         * Opening of the broad ligament via round ligament division and ligation.
         * Gentle dissection of the bladder from the uterus was performed from lateral aspect to medially.
         * Bilateral uterine artery clamping at below the placental bed
         * Continue gentle dissection the remaining adherent part of the urinary bladder
         * Gentle attempt to delierve the placenta by gentle traction on clamp.
         * If the placenta was delievered, bilateral uterine artery ligation at multiple levels and multiple square compression sutures (if needed) to control pacental bleeding bed .
         * If the placenta was not delievered we did segmental ressection of lower uterine segment including the placenta. The affected area, once excised can be repaired and the patient was treated as though she had a classical cesarean delivery.
         * Intraperitoneal drain was inserted for early detection of intraperitoneal hemorrhage or urine leak in case of cystotomy repair or possible ureteric injury.
         * The amount of blood loss within 24 h after surgery was measured by the weight of blood-soaked disposable hip pads minus its own weight.
         * Transfusion must include not only packed red blood cells (PRBC), but also fresh frozen plasma and/or cryoprecipitate to maintain in a 2:1 ratio to prevent dillutional coagulopathy

      Outcome variables:
      1. Demographic data e.g age, parity, body mass index (BMI).
      2. Amount of blood loss by measuring Hb preoperatively and after blood transfusion.
      3. Amount of blood loss intraoperative via amount and number of tampons used.
      4. Amount of blood and blood products transfusion.
      5. Hemeostasis and analegesia postoperatively.
      6. Duration of ambulation and audible intestinal sounds.
      7. Follow up of nishe at placental bed after 6 weeks via color Doppler Ultrasoumd.
      8. Intraoperative complications e.g urinary bladder injury, ureteric injury.
      9. Postoperative complications e.g ileus, sepsis.
      10. Need for conversion to hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* 1- Age between 20 - 40 years old. 2- Gestational age between 28 - 38 weeks. 3- Any patient diagnosed as placenta previa with ultrasound criteria of accretion.

  * Criteria of accretion by Colour Doppler ultrasound include: (Berkley et al., 2013).

    1. The presence of irregular shaped placental lacunae within the placenta.
    2. Thinning of myometrium overlying the placenta.
    3. Absence of retroplacental 'non-lucent line'.
    4. Protrusion of the placenta into the bladder.
    5. Increased vascularity of the uterine serosa-bladder interface.
    6. Turbulent blood flow through the lacunae on Doppler ultrasonography.

       Exclusion Criteria:

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Outcome variables: Need for conversion to hysterectomy. | 30- 90 minutes
  control of bleeding and need for removal of uterus.
Blood Loss. | During operation and 24 hours postpartum.
  Amount of blood loss ,Number of packed red blood cells and blood products transfusion.

SECONDARY OUTCOMES:
Intraoperative complications | During operation and postpartum period.
  urinary bladder injury, ureteric injury. Postoperative complications e.g ileus, sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Hamed E Ellakwa, Study Director — Menoufia
Locations (2):
- Egypt (2):
  - Menoufia University hospital, Shibīn al Kawm, Menoufia
  - Hamed Elsayed Ellakwa, Shibīn al Kawm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elkhouly NI, Solyman AE, Anter ME, Sanad ZF, El Ghazaly AN, Ellakwa HE. A new conservative surgical approach for placenta accreta spectrum in a low-resource setting. J Matern Fetal Neonatal Med. 2022 Aug;35(16):3076-3082. doi: 10.1080/14767058.2020.1808616. Epub 2020 Aug 25. PMID 32842821